CLINICAL TRIAL: NCT06006052
Title: Evaluation of Demineralized Dentin Matrix as a Scaffold for Revascularization in Immature Permanent Incisors: A Randomized Controlled Trial and an In -Vitro Study
Brief Title: Regenerative Endodontic in Immature Permanent Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Abozed mahmoud, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AnishamsU ASU
Record Dates: First submitted 2023-07-30; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Dental Trauma
MeSH Terms: interventions — Regenerative Endodontics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- study group DDM (Experimental): Group I: 10 teeth will be treated with demineralized dentin matrix attached to collagen membrane as a scaffold in the regenerative endodontic procedure.
  Interventions: Combination Product: regeneration technique
- Control group (Active Comparator): Group II: 10 teeth will be treated with the conventional regenerative endodontic procedure (blood clot scaffold).
  Interventions: Combination Product: regeneration technique
- positive control (Active Comparator): Group III: 10 teeth will be treated with collage membrane as a scaffold in the regenerative endodontic procedure
  Interventions: Combination Product: regeneration technique

INTERVENTIONS:
Combination Product: regeneration technique — clinical procedure of regenerative endodontic as AAE mentioned using different material in each group
  Other Names: regenerative endodontic

SUMMARY:
Compare the clinical and radiographic outcomes of demineralized dentin matrix scaffold to blood clot scaffold in immature permanent incisors with non-vital pulps for one year (in vivo).

Investigate the effect of demineralized dentin matrix (DDM) on dental pulp stem cells (DPSCs) (in vitro).

DETAILED DESCRIPTION:
Necrosis of the immature pulp not only is one of the multiple factors affecting long-term tooth endurance and preservation but also can act as a source of bacterial infection in the periapical area and even the maxillofacial spaces

* The use of regenerative endodontic techniques (RET) have gained popularity in the past decade with several endodontic and pediatric dentistry organization recognizing this technique as a viable technique for immature permanent teeth with necrotic pulps Regenerative endodontics are defined as biologically based techniques planned to physiologically replace impaired tooth structure, including dentin and root constructions, as well as cells of the pulp-dentin complex
* They offer the benefit of root lengthening, thickening, and subsequent apical closure which is not achievable with conventional nonsurgical endodontic treatment (NSET). The success rate of the blood clot (RET) in immature teeth has been reported to be 97.8% .The American Association of Endodontists and the European Society of Endodontology developed evidence-based protocols. To help reduce some of the differences in the RET steps such as EDTA ethylene diamine tetra acetic acid and sodium hypochlorite use, however, variations in terms of intracanal medicament, scaffold, and assessment tools still exist due to the lack of high-quality evidence

A fundamental component of the regenerative endodontic process is the presence of a scaffold for stem cells from the apical papilla to adhere, multiply and differentiate. Based on the results of many studies, the use of blood clot Regenerative procedure is not considered a true scaffold system. But it is an essential part of any appropriately designed tissue engineering regenerative endodontic strategy

.

Different treatment options and scaffolds have been tested in regenerative endodontics. Only

some of them exhibited clinical relevance such as blood clot, platelet-rich plasma, and platelet- rich fibrin as RET scaffolds. Therefore, the use of a suitable scaffold is an essential part of tissue

engineering regenerative endodontic strategy .

Hence, developing a new dental material that retains the proteins or factors that can stimulate regenerative processes close to the natural process seems promising . Tissue-derived extracellular matrices have recently been known as naturally-derived scaffolds for tissue regeneration in various applications and have been revealed to serve as a cultural substrate on which cells tend to adhere to and proliferate well and can induce regeneration specific to tissues and sites

A new extracellular matrix material, demineralized dentin matrix (DDM) derived from extracted teeth has been found to act as a biocompatible scaffold for the attachment, differentiation, and proliferation of human DPSCs (dental pulp stem cell) into odontoblast-like cells . The dentin matrix has proposed roles for directing mineralized tissue repair in dentine and bone; however, the range of bioactive components in dentine and specific biological effects on bone-derived mesenchymal stem cells (MSCs) in humans are less well understood

.

DDM is an autogenous tooth dentin that has osteoconductive and osteoinductive potential since it contains extracellular collagen-1 and various growth factors. DDM as a solid blocky material has less physical stability and sealing ability as a material for regenerative endodontics.

Therefore it has been further fabricated into the forms of DDM powder, gel, and sheets to maintain bioactivity .

DDM can be prepared with low risks of infection and rejection with noninvasive attainability; thus, it should be considered a natural resource to be used to full advantage for other applications

indicated that DDM as a regenerative biomaterial has potential roles in tissue regeneration. However, to confirm these trials, further well-designed analyses are needed, and an evaluation of adverse events in observational studies is also needed. To our knowledge, DDM has not been investigated as a scaffold in regenerative endodontics for permanent teeth. Several studies evaluated the regenerative effect of DDM on the dentin-pulp complex through the direct pulp capping technique, and it was found to possess the ability to activate the odontogenic differentiation of stem cells resident in the pulp tissues and induce reparative dentin formation. DDM is also considered for the alveolar ridge, maxillary sinus floor augmentations, socket preservation, furcation perforation repair, guided bone, and bio root regenerations as well as bone and cartilage healing

.

Hence, this study will be designed to evaluate the regenerative effect of Demineralized Dentin Matrix as a scaffold in comparison to a conventional blood clot in immature permanent teeth.

ELIGIBILITY:
Inclusion Criteria : patients clinical examination Must be include the following

* Patients aged 7-13years at the time of enrolment.
* Provision of informed consent by one parent or legal guardian.
* At least the patents have one immature permanent anterior tooth diagnosed with irreversible pulpitis or pulp necrosis with or without periapical lesions.
* Restorable teeth ,clinical crown should be enough to use rapper dam Compliant patient/parent.
* Patients are not allergic to medicaments and antibiotics necessary to complete the procedure (ASA 1 or 2).
* Radiologic evidence of open apices (Teeth are considered immature when a minimum of 0.8 mm apical foramen width is evident)
* Exclusion Criteria:
* the patients will excluded if one of the following criteria is present in the patients
* Teeth with root fractures.
* Presence of internal or external root resorptions.
* Developmental anomalies of the root.
* Presence of periapical radiolucency more than 10 mm.
* Tooth with class III mobility.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
the elimination of symptoms at base line at 0,3 and 6 and 9and 12 month | at 0,3 and 6 and 9and 12 month
  no history of pain, using Visual Analog Score for pain, measure quality of life.
  soft tissue swelling or sinus tract by visual examination , Sensitivity to percussion, Tooth mobility by clinical assessment by operator

SECONDARY OUTCOMES:
change root wall thickness and root length in radiographic measurement in millimeter at 0,3,6,9,12 month | at 0, 3 and 6 and 9and 12 month
  change root length and width measured in mml by digital radiography using parallel technique

OTHER OUTCOMES:
change root wall thickness and root length using CBCT millimeter at base line and after 12 month | at base line and after 12 month
  cone beam computed tomography using OnDemand soft wear and measure the 3d tooth root wall thickness and root length

CONTACTS AND LOCATIONS:
Overall Officials: nagwa khattab, professor, Study Director — Ain Shams University
Locations (1):
- Ain shams university, Cairo, Alabbassia, Egypt

IPD SHARING:
Plan to Share IPD: No
regeneration immature teeth

REFERENCES:
- See also: Regeneration of Tooth with Allogenous, Autoclaved Treated Dentin Matrix with Dental Pulpal Stem Cells: An In Vivo Study — https://doi.org/10.1016/j.joen.2020.05.016

DOCUMENTS (1):
  • Study Protocol (2023-07-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT06006052/Prot_000.pdf